CLINICAL TRIAL: NCT07174661
Title: Empowerment Through Preparedness: Improving Advance Care Planning (ACP) in Adolescents and Young Adults (AYAs) With Advanced Solid Malignancies and High-Grade Brain Tumors
Brief Title: Educational Tools for the Improvement of Early Advance Care Planning in Adolescents and Young Adults With Advanced Solid Tumors and High-Grade Brain Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-007280; NCI-2025-06307 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-007280 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Neoplasm; Malignant Brain Neoplasm; Recurrent Advanced Malignant Solid Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Advance Care Planning; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (early ACP) (Experimental): Patients watch a brief, on-demand early ACP educational video at baseline and then one month later attend an ACP appointment with either an AYA social worker or AYA palliative medicine physician assistant over 1 hour.
  Interventions: Behavioral: Advance Care Planning; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Behavioral: Advance Care Planning — Attend ACP appointment
Other: Educational Intervention — Watch on-demand early ACP educational video
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Electronic Health Record Review — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies whether educational tools work to improve early advance care planning (ACP) in adolescents and young adults (AYAs) with solid tumors that may have spread from where they first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) and high-grade brain tumors. The incidence of AYA cancers is on the rise with approximately 90,000 new diagnoses yearly in the United States. Cancer remains the leading cause of disease-related death among AYAs, which could be due to patients having more advanced disease at presentation. It is recommended that AYAs begin ACP conversations at the start of treatment. ACP includes clarifying goals of care, discussions about end-of-life preferences, and completing a legal document that states the treatment or care a person wishes to receive or not receive if they become unable to make medical decisions (advance directive). The educational tools in this study include an early ACP educational video featuring AYAs with cancer and an ACP appointment geared for AYAs. Patients can access and watch the educational video at home prior to their scheduled ACP appointment. During the ACP appointment, a tailored ACP guide made specifically for AYAs is reviewed and questions regarding ACP are answered. This may help to introduce the importance of key ACP concepts, which may improve early ACP in AYAs with advanced solid tumors and high-grade brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39 at initial cancer diagnosis

  * Patient <18 years of age are not included in this pilot as Mayo Clinic in Arizona (MCA) does not treat pediatric patients
* Recently diagnosed (defined as 12 months or less from initial diagnosis or advance stage relapse) with either a stage III/IV solid malignancy or high-grade brain tumor. This includes patients who have stage III/IV recurrence of previously stage I/II solid malignancy
* Actively receiving primary oncologic care at Mayo Clinic Arizona
* Able to read, understand, and speak English
* Those who have completed prior advance directive documents are still eligible to participate.

Exclusion Criteria:

* Age < 18 or > 39 at initial cancer diagnosis
* Diagnosed with stage I/II solid malignancy, low-grade brain tumor, or hematologic malignancy
* Not receiving primary oncologic care at Mayo Clinic Arizona
* Unable to read, understand, and speak English
* Patients > 12 months from initial diagnosis or advanced stage relapses, in survivorship or on hospice
* No internet or computer/smart phone access

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing routine, early Advance Care Planning (ACP) | Up to 1 year
  Feasibility is achieved if 60% of participants can complete the baseline survey, view the pre-appointment educational video, and attend the hour-long ACP appointment. Baseline survey completion will be defined as answering at least 80% of the survey questions. Video viewing will be assessed via a single yes/no survey item presented after the video. Results will be analyzed descriptively.
Satisfaction with each intervention component (Acceptability) | Up to 1 year
  Acceptability is defined as majority satisfaction with each intervention component. Participants will be asked to rate their experience with the educational ACP video and ACP appointment on a 4-point Likert scale (e.g., very helpful, somewhat helpful, a little helpful, not helpful) using 4 questions regarding each intervention's usefulness and recommendations to peers. Higher scores indicate greater satisfaction and/or greater likelihood of recommending to peers. Descriptive statistics will be utilized to broadly analyze the sample.

SECONDARY OUTCOMES:
Advance directive completion rates | Up to 1 year
  Assess by review of medical record to determine whether there was an increase in advance directive completion rates within the electronic medical record, as compared to historical institutional records (control). Descriptive statistics will be utilized to broadly analyze the sample.
Change in ACP readiness | Baseline; 4 months; 7 months
  Assessed using 4 validated multiple-choice questions. Scores range from 0-20, with higher scores indicating increased readiness. In patients indicating that they signed official advance directive paperwork, an additional yes/no question will be asked to assess if any updates were made to advance directive documents (i.e. living will or surrogate decision maker/medical power of attorney) since that time. A mixed linear effect model will be used to analyze longitudinal changes.
Change in ACP anxiety | Baseline; 4 months; 7 months
  Assessed using a single question on a 4-point Likert scale. A mixed linear effect model will be used to analyze longitudinal changes.

CONTACTS AND LOCATIONS:
Overall Officials: Allison C. Rosenthal, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials